CLINICAL TRIAL: NCT05888441
Title: Impact of Stepping Over Obstacles of Different Contrast and Height on Gait and Eye Movements in Older Adults With and Without Vision Impairment
Brief Title: Obstacle Negotiation in Older People With and Without Vision Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Shirin E. Hassan, Associate Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16447
Record Dates: First submitted 2023-05-04; First posted 2023-06-05 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Low Vision
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Vision Group (Experimental): At a single study visit, the group of low vision participants will be asked to perform a series of short walking trials. During each trial they will walk at a self-selected speed along a walkway (6 meters in length) that may or may not contain an obstacle to step over. The trials will be randomly varied with regard to an obstacle's presence, height, and contrast from the walkway surface. Repeated trials of each condition variation will be performed during the visit.
  Interventions: Other: Obstacle characteristics
- Control Group (Active Comparator): At a single study visit, the group of age-matched participants without low vision will be asked to perform a series of short walking trials. During each trial they will walk at a self-selected speed along a walkway (6 meters in length) that may or may not contain an obstacle to step over. The trials will be randomly varied with regard to an obstacle's presence, height, and contrast from the walkway surface. Repeated trials of each condition variation will be performed during the visit.
  Interventions: Other: Obstacle characteristics

INTERVENTIONS:
Other: Obstacle characteristics — In the walking trials, when an obstacle is present, the obstacle height and obstacle contrast level will be varied across the trial repetitions.
  Each participant will be exposed to obstacles of two heights: the first will be 1 centimeter in height, and the second will be approximately 20% of the subject's leg length (ranging in physical height between 15 - 22 centimeters to cover a range of leg lengths in the population).
  Obstacles (of both heights) will also be painted such that their measured luminance (or contrast) level against the floor luminance is varied. High contrast obstacles will have ≥80% Michelson contrast and low contrast obstacles will have ≤30% Michelson contrast.

SUMMARY:
Falls are common among people with vision impairment and can lead to devastating health consequences. Understanding the functions of vision and how the visual characteristics of obstacles in the walking path impact the gait of people with vision impairment is necessary to create strategies to prevent falls in this population. The purpose of this study is to determine how adults with vision impairment change their gait behavior when stepping over obstacles that vary in height and contrast to the ground. We will then determine the mechanisms of gaze behavior that correlate to the gait behavior.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Able to walk independently
* Either have normal vision, or impaired vision.

  * Impaired vision is defined as binocular visual acuity of 20/25 or worse with or without a central scotoma; and/or binocular visual field that is restricted to an average of 100 degrees in diameter or less
  * Control subjects will have visual acuity of 20/40 or better.

Exclusion Criteria:

* Not cleared by a medical provider for moderate physical activity
* Self-report or have a history of: vestibular disorder or deafness
* Medical history of any condition that affects the ability to walk for up to 2 hours with breaks, such as feeling dizzy or faint, chest pain, palpitations, pain or numbness in the legs, shortness of breath,
* Cognitive limitations either by self-report or a score on the Mini Mental State Exam below 24 (out of 30)
* Walking or gait abnormalities, such as those caused from an injury, surgery, severe arthritis, or neurological condition such as Parkinson's disease
* Unable to walk without any walking aids such as a walker, cane, guide dog, or oxygen tank.
* Does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Vertical foot clearance, lead limb | During a single intervention visit (Study Visit 2), up to 2-3 hours in duration.
  Distance from lowest point of foot (heel or toe) to top of obstacle
Foot placement variability | During a single intervention visit (Study Visit 2), up to 2-3 hours in duration.
  Standard deviation of position of toe to obstacle over 2-4 steps before the obstacle
Obstacle crossing speed | During a single intervention visit (Study Visit 2), up to 2-3 hours in duration.
  Speed from lead toe off immediately before the obstacle to trail heel down immediately after the obstacle.
Gaze sequencing | During a single intervention visit (Study Visit 2), up to 2-3 hours in duration.
  Sequence of fixations from start of trial to end of trial, normalized to the total duration and divided into 100 equal segments

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No